CLINICAL TRIAL: NCT04693026
Title: Efficacy of Ramdicivir and Baricitinib Combination Therapy for the Treatment of COVID 19 ARDS
Brief Title: Efficacy of Ramdicivir and Baricitinib for the Treatment of Severe COVID 19 Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: M Abdur Rahim Medical College and Hospital (Other Government)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Abu Taiub Mohammed Mohiuddin Chowdhury, Resident, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M.A.R.M.C.D./2020/2637
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Covid-19 ARDS
Keywords: COVID 19; Covid-19 ARDS; Tocilizumab; Remdicivir; Baricitinib
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; baricitinib; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Remdesivir + Baricitinib treatment group (Experimental): Remdesivir (Injectable solution):
  A loading dose of Remdesivir I/V 5mg/kg (less than 40kg) or 200mg (>40kg) on day 1, then 2.5mg/kg (less than 40kg) or 100mg (>40kg) daily following randomization.
  +
  Baricitinib (oral tablet form):
  Baricitinib tablets 4 mg/day for 2 to 4weeks
  Interventions: Drug: Remdesivir; Drug: Baricitinib
- Group B: Remdesivir + Tocilizumab treatment group (Active Comparator): Remdesivir (Injectable solution) A loading dose of Remdesivir I/V 5mg/kg (less than 40kg) or 200mg (>40kg) on day 1, then 2.5mg/kg (less than 40kg) or 100mg (>40kg) daily following randomization.
  +
  Tocilizumab (Injectable solution):
  Tocilizumab I/V 8mg/Kg up to 800mg highest 12 hours apart.
  Interventions: Drug: Remdesivir; Drug: Tocilizumab

INTERVENTIONS:
Drug: Remdesivir — Remdesivir 100 IV Infusion as a lyophilized powder
  Other Names: Ninavir
Drug: Baricitinib — Baricitinib oral tablet form
  Arms: Group A: Remdesivir + Baricitinib treatment group
Drug: Tocilizumab — Tocilizumab IV Infusion
  Arms: Group B: Remdesivir + Tocilizumab treatment group

SUMMARY:
This study was designed to evaluate the efficacy of Remdesivir and Baricitinib combination therapy for the treatment of severe Acute Respiratory Distress Syndrome (ARDS) caused by Coronavirus disease 2019 (COVID-19). Our aim is to compare the outcome of the "Remdesivir + Baricitinib" combination against "Remdesivir + Tocilizumab" therapy and find the best option for the management of ARDS in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

Severe COVID-19 patients require hospitalization under HDU/ICU. The SARSCoV-2 infection will be confirmed by RT PCR / CT Chest in every case.

Exclusion Criteria:

Participants with uncontrolled clinical status who were hospitalized from the before. Contraindication / possible drug interaction. Participants who have any severe and/or uncontrolled medical conditions like, Severe ischemic heart disease, epilepsy, malignancy, Pulmonary/ renal/hepatic disease, AIDS, Pulmonary TB, pregnancy, Corpulmonale, and etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-03-05 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Improvement (TTCI) | Following randomization 30 days
  Time to Clinical Improvement (TTCI) Defined as Time from Randomization to National Early Warning Score 2 (NEWS2) Score of </= 2 Maintained for 24 Hours.

SECONDARY OUTCOMES:
Mortality Rate | Following randomization 30 days.
  Mortality Rate on Days during hospitalization
Duration of ICU stay | Following randomization 30 days.
  Duration of ICU Stay in days.
Duration total hospital stay | Following randomization 30 days.
  Duration of hospital stay in days.
Rate of daily Supplemental Oxygen Use | Following randomization 30 days.
  Rate of daily Supplemental Oxygen Use by the patient
Time to Clinical Failure | Following randomization 30 days.
  Time to Clinical Failure, Defined as the Time from Randomization to the First Occurrence of Death, Mechanical Ventilation, ICU Admission, or Withdrawal (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Abu Taiub Mohammed Mohiuddin Chowdhury, MBBS, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University; Akter Kamal, MD, PhD, Study Director — M Abdur Rahim Medical College and Hospital
Locations (1):
- M. Abdur Rahim Medical College Hospital, Dinajpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No